CLINICAL TRIAL: NCT02245750
Title: Value of Routine Hysteroscopy Prior to IVF/ICSI Cycles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, mostafa fouad, Value of Routine Hysteroscopy prior to IVF/ICSI Cycles: A Randomized Control Trial, Ain Shams Maternity Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Routine Hysterscopy
Record Dates: First submitted 2014-04-24; First posted 2014-09-22 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Infertility
Keywords: hysteroscopy - recurrent implantation failure
MeSH Terms: conditions — Infertility | interventions — Hysteroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Routine Invistigations (No Intervention): ICSI with long luteal phase protocol
- Hysteroscopy (Experimental): hysteroscopy will be done prior to the ICSI cycle
  Interventions: Device: Hysteroscopy

INTERVENTIONS:
Device: Hysteroscopy — hysteroscopy and endometrial injury prior to the IVF/ICSI cycle
  Arms: Hysteroscopy

SUMMARY:
In the current study the investigators hypothesize that Routine Hysteroscopy prior to IVF/ICSI cycle increases the clinical pregnancy rate.

DETAILED DESCRIPTION:
A randomized controlled study involving 300 patients with recurrent implantation failure

ELIGIBILITY:
Inclusion Criteria:

1. Patient's age ranged from 20-40 years.
2. Normal appearance of the uterine cavity on hysterosalpingography.
3. Patients prepared for IVF/ICSI cycle.

Exclusion Criteria:

1. Patients who have any contraindications for hysteroscopy. (Menstruation, pregnancy, severe vaginitis or cervicitis, endometrial infection and history of Pelvic Inflammatory Diseases).
2. Patients with uterine cavity pathology previously known to the examiner.
3. Patients with previous uterine surgery such as myomectomy.
4. Patients with abnormal HSG.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-08; Primary Completion 2014-12 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
• Clinical pregnancy rate. | 6 months

SECONDARY OUTCOMES:
• Live Birth Rate | 6 months

OTHER OUTCOMES:
• Uterine anomalies detected by Hysteroscopy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: mostafa f gomaa, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams Maternity hospital, Cairo, Egypt